CLINICAL TRIAL: NCT04672642
Title: Evaluation of the SpyGlass DS vs Standard Method for Detection of Residual Pancreatic Calculations After Endoscopic Treatment
Brief Title: Evaluation of the SpyGlass DS for Detection of Residual Pancreatic Calculations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SPY PCC 2020
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2021-07

CONDITIONS: Pancreatitis, Chronic
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SpyGlass DS after endoscopic treatment (Experimental)
  Interventions: Device: SpyGlass DS

INTERVENTIONS:
Device: SpyGlass DS — Detection by the SpyGlass DS of residual pancreatic stones not detected by the standard method (CT scan and ERCP)

SUMMARY:
The purpose of the study is to assess the efficacy of the SpyGlass DS for the detection of residual pancreatic calculations after endoscopic treatment.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 and over;
* with chronic calcifying pancreatitis;
* having already received endoscopic treatment for pancreatic pain related to stenosis and / or pancreatic stones;
* having given free, informed and written consent;
* being affiliated to a social security scheme or beneficiary of such a scheme.

Exclusion Criteria:

* contraindications to performing an upper digestive endoscopy;
* haemorrhagic disease, haemostasis and coagulation disorder (PR <60%, PTT> 40 s and platelets <60,000 / mm3;
* pregnant or breastfeeding woman;
* adult patient protected (guardianship or curatorship), or deprived of liberty by a judicial or administrative decision;
* person subject to a safeguard measure.

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
Residual pancreatic stones detected by the Spyglass DS | baseline
  rate of residual pancreatic stones detected by the SpyGlass DS, after a treatment by CT-scan and ERCP (recommended standard method) showing no stones in the Wirsung's duct. .

SECONDARY OUTCOMES:
Residual pancreatic stones extracted by the SpyGlass DS accessory (the SpyGlass Basket) | baseline
  rate of residual pancreatic stones extracted by by the SpyGlass DS accessory (the SpyGlass Basket) after being detected by the SpyGlass DS.
VAS score for pancreatic pain | preoperative, 1 month, 6 months and 12 months
  pain visual analogue scale from 0 (no pain) to 10 (worst pain possible)
Analgesic consumption | preoperative, 1 month, 6 months and 12 months
  level of analgesic (if several analgesics of different levels are used, the analgesic of the highest level will be taken into account each time)
Analgesic consumption | preoperative, 1 month, 6 months and 12 months
  total daily dose (mg)
Rate of patients hospitalized for pancreatic pain | 12 months
Rate of operated patients requiring partial / total pancreatectomy, or pancreas-jejunal shunts for pancreatic pain | 12 months
Rate of patients requiring endoscopic treatment (placement of pancreatic-duct stent, extraction of pancreatic stones) | 12 months
Self-administered quality of life questionnaire score | preoperative, 1 month, 6 months and 12 months
  36-Item Short Form Health Survey (SF-36). SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. A score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
AE rate and type | during and immediately after the operation, 7 days, 1 month, 6 months and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Saint Jospeh Marseille, Marseille, France